CLINICAL TRIAL: NCT06529588
Title: Soluble Urokinase Plasminogen Activator Receptor (suPAR) is a Potential Biomarker of Stage III-IV, Grade C Periodontitis Through the Impact of Post-radiotherapy on Head and Neck Cancer Patients
Brief Title: Estimation of (suPAR) in Chronic Periodontitis With Post-radiotherapy on HNCs Patients
Acronym: HNCs
Status: Completed | Type: Observational
Sponsor: Al-Maarif University College (Other)
Responsible Party: Sponsor
Other Study IDs: suPAR as a potential biomarker
Record Dates: First submitted 2024-06-18; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Cancer; Chronic Periodontitis; Radiotherapy Side Effect
Keywords: Chronic Periodontitis; Head and Neck Cancer; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Chronic Periodontitis; Radiation Injuries | interventions — Radiation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer post-radiotherapy: Head and Neck cancer patients who received radiotherapy (32-35 fractions) exposure (5700-7000 Gys) addition chemotherapy (cisplatin or cetuximab (2-3 dosages).
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — HNCs patients who received radiotherapy was exposure (5700-7000 Gys) for fractions number (32-35) after 6 months
  Other Names: Head and neck cancer patients after 6 irradiation

SUMMARY:
This study aims to improve a soluble urokinase plasminogen activator receptor suPAR is a reliable biomarker of chronic periodontitis and may be replaced in patients with head and neck cancer post-radiotherapy (HNC post-RT).

DETAILED DESCRIPTION:
The urokinase-type plasminogen activator receptor (uPAR) plays an essential function in leukocytes and endothelial homeostasis and, therefore, in the development of chronic periodontitis. The study enrolled 150 participants, 50 chronic periodontitis with head and neck cancer post radiotherapy (CP+HNC post-RT) patients, 50 chronic periodontitis (CP) without HNC patients, and 50 healthy controls. Clinical Attachment Loss (CAL), Probing Pocket Depth (PPD), Plaque Index (PI), and Gingival Bleeding Index (GBI) were recorded. An enzyme-linked immunosorbent assay (ELISA) was constructed to quantify serum (suPAR) levels.

ELIGIBILITY:
Inclusion Criteria:

* A pathologically confirmed malignant neoplasm of HNC (derived from epithelial cells).
* Not having received radiation therapy previously.
* No distant metastasis.
* No history of salivary gland surgery (parotid, submandibular, or sublingual).
* A generally satisfactory physical condition with a performance score of 0 to 1 point and a planned survival period of more than a year and scores of 2 higher indicating increasing disability.

Exclusion Criteria:

* Previous oral disease or salivary gland disease history.
* Definitive diagnosis of multiple sclerosis, xerostomia, or systemic disease.
* Refusal to participate in the study.

Ages: 28 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study was n=26 nasopharyngeal tumors (n=20 nonkeratinizing and n=6 keratinizing carcinomas), (n=6 oropharyngeal squamous cell carcinoma, SCC), (n=8 Laryngeal cancer), (n=6 tongue cancer), and (n=4 primary malignancies of unclear origin). Twenty-eight of the patients (or 56%) had a concomitant systemic therapy (2-3 doses) of cisplatin or cetuximab in addition to radiotherapy. Chronic periodontitis patients without HNCs included: Patients' average ages ranged from 28 to 65 years, with 40 (80%) of them being male. More than half of them had a history of smoking, with 31 (62%) and 5 (10) of them having used alcohol. A control group was used periodontally healthy as a controlled study, the mean age was 40.12 years (min-max: 29-60 years).
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Measure of serum suPAR level | 6 months
  Measure of serum suPAR level in patients head and neck cancer who received radiotherapy
Clinical Periodontal parameters measured | 6 months
  Periodontal parameters included (CAL, PI, GBI, PPD) measured by using a millimeter periodontal probe in patients with head and neck cancer who received radiotherapy.

SECONDARY OUTCOMES:
Oral pH-saliva was measured | 6 month
  Oral pH-saliva collected from outcomes and measured pH-saliva by using pH-meter in patients who underwent radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Al-Kubaisi, PhD, Study Director — Al-Maarif University College
Locations (1):
- Ahmed A. Al-Kubaisi, Ramadi, Al-Anbar Governorate, Iraq

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lalla RV, Treister NS, Sollecito TP, Schmidt BL, Patton LL, Helgeson ES, Lin A, Rybczyk C, Dowsett R, Hegde U, Boyd TS, Duplinsky TG, Brennan MT. Radiation therapy for head and neck cancer leads to gingival recession associated with dental caries. Oral Surg Oral Med Oral Pathol Oral Radiol. 2022 May;133(5):539-546. doi: 10.1016/j.oooo.2022.01.016. Epub 2022 Jan 31. PMID 35304084
- [Result] Gasparoni LM, Alves FA, Holzhausen M, Pannuti CM, Serpa MS. Periodontitis as a risk factor for head and neck cancer. Med Oral Patol Oral Cir Bucal. 2021 Jul 1;26(4):e430-e436. doi: 10.4317/medoral.24270. PMID 33340075
- [Derived] Al-Kubaisi AA, Ghazi MA, Majeed NS, Aldelaimi ER, Enezei HH. Soluble urokinase plasminogen activator receptor (suPAR) is a potential biomarker of stage III-IV, grade C periodontitis through the impact of post-radiotherapy on head and neck cancer patients. BMC Oral Health. 2024 Sep 27;24(1):1144. doi: 10.1186/s12903-024-04801-w. PMID 39334335